CLINICAL TRIAL: NCT02342821
Title: Empowering Immigrants in the Greater Boston Area to Connect to HBV Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Fusco, Dahlene N.,M.D.,Ph.D., Physician, Massachusetts General Hospital
Other Study IDs: IN-US-174-1254
Record Dates: First submitted 2015-01-16; First posted 2015-01-21 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This Study will attempt to provide information / linkage to HBV care for persons at risk in the Greater Boston area.

DETAILED DESCRIPTION:
Specific Aims

1. Provide HBV education at community sites where immigrants at risk for HBV could be informed of the risks related to HBV, in a culturally and linguistically sensitive manner.

   1. Chelsea, Charlestown, and Revere MGH Community Health Centers: posters, pamphlets, and telephone line to provide HBV education
   2. Senegalese Community Center: community meeting, posters, and pamphlets
   3. African Students' Association, Suffolk University: community meeting, posters, and pamphlets
   4. Revere Cambodian Community Centers: community meeting, posters, and pamphlets
2. Provide at-risk persons with the tools to develop an HBV diagnosis plan with his / her provider.

   1. Provide counseling on the significance of different testing results prior to testing
   2. Connect to testing, and appropriate post-test follow-up appointments
3. Provide an education hub for patients and providers to return to with questions regarding: test interpretation, available treatments for those who test positive, and screening for hepatocellular carcinoma in those who are infected.

   1. Provide copy of an easy to understand US HBV treatment algorithm in native languages
   2. Provide information related to genotype-specific risks for HCC (increased with GT C).

ELIGIBILITY:
Inclusion Criteria: all persons interested in hearing more information about HBV -

Exclusion Criteria: children

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: immigrants and other persons at HBV risk in Greater Boston area
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Improved understanding of HBV by Questionnaire | 1 year
  Participants will be provided questionnaires by D. Fusco